CLINICAL TRIAL: NCT04558697
Title: Use of Vagitories Based on St. John's Wort, Tea Tree Oil and Shepherd's Purse in the Treatment of Vaginal Inflammation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sarajevo (Other)
Collaborators: Institution for Health Protection of Women and Motherhood (Unknown); University of Tuzla (Unknown)
Responsible Party: Principal Investigator, Kemal Durić, PhD, Kemal Duric PhD, Associate Professor, University of Sarajevo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03/7-1053/19
Record Dates: First submitted 2020-08-31; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Non Specific Vaginitis
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Shepherd's Purse extractum oleosum vagitories (Experimental): Vagitories containing Calendulae extractum oleosum 5,5% (w/w), Bursae pastoris extractum oleosum 5,5% (w/w), Matricariae extractum oleosum 5,5% (w/w), Hyperici extractum oleosum 5,5% (w/w) and Millefolii extractum oleosum 5,5% (w/w) as active component
  Interventions: Drug: Shepherd's Purse extractum oleosum vagitories
- Tea tree oil vagitories (Experimental): Vagitories containing tea tree oil, 200 mg per each vagitorie as active component
  Interventions: Drug: Tea tree oil vagitories
- Hyperici extractum oleosum vagitories (Experimental): Vagitories containing Hyperici extractum oleosum 32% (w/w) as active component
  Interventions: Drug: Hyperici extractum oleosum vagitories
- Vagitories - Probiotic (Active Comparator): Commercially available vagitories with probiotic
  Interventions: Drug: Vagitories - Probiotic

INTERVENTIONS:
Drug: Shepherd's Purse extractum oleosum vagitories — Shepherd's Purse extractum oleosum vagitories will be administered once daily for 5 days
  Arms: Shepherd's Purse extractum oleosum vagitories
Drug: Tea tree oil vagitories — Tea tree oil vagitories will be administered once daily for 5 days
  Arms: Tea tree oil vagitories
Drug: Hyperici extractum oleosum vagitories — Hyperici extractum oleosum vagitories will be administered once daily for 5 days
  Arms: Hyperici extractum oleosum vagitories
Drug: Vagitories - Probiotic — Vagitories - Probiotic will be administered once daily for 5 days
  Arms: Vagitories - Probiotic

SUMMARY:
There are more and more herbal preparations that are used for the purpose of treatment and improvement of the clinical picture of vaginitis by patients themselves, but also by healthcare professionals. Plant species, St. John's wort, chamomile, calendula, yarrow, shepherd's purse and tea tree oil are well known for there anti-inflammatory, antimicrobial and wound healing activity. This paper presents the results of a clinical study in which three herbal formulations/vagitories, based on extracts of above mentioned plant species, were investigated for their effectiveness on non-specific vaginitis.

This was randomized controlled clinical study that included 210 women with diagnosed non-specific vaginitis. Patients were divided into two basic groups, women in reproductive stage and postmenopausal stage. Three subgroups, containing approximately 30 patients each, received one of three vagitorie formulations for 5 days during which the effects on subjective and objective symptoms were monitored.

ELIGIBILITY:
Inclusion Criteria:

* adult women who already had sexual intercourse
* diagnosis of non-specific vaginal inflammation by medical examination.

Exclusion Criteria:

* microbiologically confirmed bacterial vaginosis,
* treatment with antibiotic therapy according to official protocols and guidelines
* allergies to one of the plant species included in the vaginal test,
* diabetes mellitus,
* pregnancy,
* lactation,
* immunodeficiency disorder,
* severe chronic illness,
* previous radiotherapy, chemotherapy and biological therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 210 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in objective symptoms of non-specific vaginitis, assessed by gynecological examination | 1 day after treatment completion
  The clinical symptoms and signs, including redness, hyper-secretion, local edema, pain and annealing were diagnosed at the baseline and 5 days after the beginning of the treatment. Gynecologist determined only the presence or absence of the above mentioned symptoms.

SECONDARY OUTCOMES:
Change in subjective symptoms of non-specific vaginitis, assessed by the valuation of subjective parameter of vaginitis reported by patients during gynecological examination | 1 day after treatment completion
  Subjective symptoms including vaginal secretion, itching and dryness of the vaginal mucous were diagnosed at the baseline and 5 days after beginning of the treatment. During anamnesis gynecologist determined the presence or absence of the above mentioned symptoms.
Incidence of vaginitis correlated with age, life habits and sexual behavior, assessed by questioner | Through study completion, an average of 3 months
  At the baseline, the patents completed a questionnaire that included questions regarding their age, life habits (permanent relationship, smoker, use of alcohol,number of births, abortion number) and sexual behavior (number of partners, years of first sexual intercourse, contraceptive use, previous presence of sexually transmitted diseases). The incidence of vaginitis correlated to above mentioned demographic data will be assessed by questioner

CONTACTS AND LOCATIONS:
Overall Officials: Fahir Becic, PhD, Study Chair — Universiyt of Sarajevo Faculty of Pharmacy
Locations (1):
- Kemal Duric, Sarajevo, Canton Sarajevo, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: No